CLINICAL TRIAL: NCT01372683
Title: The Effect of Oat Based Breakfast Cereals on Satiety
Brief Title: Oat Breakfast Satiety Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP 1103
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Subjective Appetite and Satiety; Subjective Energy Levels
Keywords: Appetite; Satiety; Subjective energy; Oats
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test cereal 1 (Experimental): Oat based breakfast cereal
  Interventions: Other: Dietary Intervention
- Test cereal 2 (Experimental): 2nd Oat based breakfast cereal
  Interventions: Other: Dietary Intervention
- Leading oat based RTE cereal (Experimental): 3rd oat based breakfast cereal
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Comparison of oat based breakfast cereals

SUMMARY:
This study is designed to test the hypothesis that on an equivalent calorie basis, oat based breakfast cereals do not provide the same satiety benefit. The study will also demonstrate the satiety comparison of the cereals related to product density.

DETAILED DESCRIPTION:
This study is designed to test the hypothesis that on an equivalent calorie basis, oat based breakfast cereals do not provide the same satiety benefit. The study will also demonstrate the satiety comparison of the cereals related to product density. Ninety-six healthy men and women 18 years of age or older will be enrolled into this study and divided into 2 groups of 48 each to investigate the satiety impact of two oat based breakfast cereals compared to the leading ready-to-eat (RTE) oat based breakfast cereal. Each subject will participate in two test sessions (1 test cereal vs the leading RTE cereal). Subjects will come to the Ingestive Behavior Laboratory between 8 and 10 am after having nothing to eat for 10 hours prior to the scheduled visit time and be given one of the three cereals. The second session will be scheduled at least 1 week after the first. Visual analogue scales of hunger, satiety and subjective energy will be completed at baseline, 30, 60, 120, 180, and 240 minutes. Subjects will return on another day separated by at least a week to repeat the breakfast. Area under the curves of appetite and satiety will be compared with a mixed model.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Healthy
* Willing to use an effective contraceptive during the study, if sexually active and capable of bearing children

Exclusion Criteria:

* Women who are pregnant or nursing
* Gain or loss of > 4kg in the last 3 months.
* Diabetes mellitus (fasting glucose >126 mg/dL)
* Dietary restraint on the Three Factor Eating Questionnaire score greater than or equal to 14
* Allergy to any of the foods used for the test breakfasts (oats or milk)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of appetite and satiety | 4 hours

SECONDARY OUTCOMES:
Area under the curve for subjective energy measures | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States